CLINICAL TRIAL: NCT06640335
Title: The Effects of Vegetable Preloading on Postprandial Glycemia, Insulinaemia and Gastric Emptying in Healthy Adults: A Randomized Cross-over Trial
Brief Title: The Effects of Vegetable Preloading on Postprandial Glycemia, Insulinaemia and Gastric Emptying
Acronym: APRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Amy Lin, PhD, Senior Principal Scientist I, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-095
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Postprandial Hyperglycemia; Insulin High
MeSH Terms: conditions — Hyperglycemia; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Control (All 24 participants) (No Intervention): Subjects consume 300 g of Russet Burbank mashed Potatoes
- Co-ingestion (All 24 participants) (Experimental): Subjects co-ingest both (300 g mashed potatoes) and (200 g baby round spinach supplemented with canola oil) in the same time.
  Interventions: Other: Co-ingestion
- 0 min preload (meal sequence) (10 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, then directly consume 300 g of mashed potatoes.
  Interventions: Other: 0 min preload
- 5 min preload (10 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 5 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: 5 min preload
- 10 min preload (10 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: 10 min preload
- 15 min preload (10 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 15 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: 15 min preload
- 20 min preload (10 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 20 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: 20 min preload
- Spinach only /10 min preload (All 24 participants) (Experimental): Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: Spinach only / 10 min preload
- (Spinach + Canola oil) 10 min preload (All 24 participants) (Experimental): Subjects consume 200 g baby round spinach WITHOUT canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: 10 min preload
- Canola oil only / 10 min preload (All 24 participants) (Experimental): Subjects consume 20 g of canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Interventions: Other: Canola oil only / 10 min preload

INTERVENTIONS:
Other: Co-ingestion — Subjects co-ingest both (300 g mashed potatoes) and (200 g baby round spinach supplemented with canola oil) in the same time.
  Arms: Co-ingestion (All 24 participants)
Other: 0 min preload — Subjects consume 200 g baby round spinach supplemented with canola oil first, then directly consume 300 g of mashed potatoes.
  Arms: 0 min preload (meal sequence) (10 participants)
Other: 5 min preload — Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 5 minutes, then consume 300 g of mashed potatoes.
  Arms: 5 min preload (10 participants)
Other: 10 min preload — Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Arms: (Spinach + Canola oil) 10 min preload (All 24 participants); 10 min preload (10 participants)
Other: 15 min preload — Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 15 minutes, then consume 300 g of mashed potatoes.
  Arms: 15 min preload (10 participants)
Other: 20 min preload — Subjects consume 200 g baby round spinach supplemented with canola oil first, wait 20 minutes, then consume 300 g of mashed potatoes.
  Arms: 20 min preload (10 participants)
Other: Spinach only / 10 min preload — Subjects consume 200 g baby round spinach WITHOUT canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Arms: Spinach only /10 min preload (All 24 participants)
Other: Canola oil only / 10 min preload — Subjects consume 20 g of canola oil first, wait 10 minutes, then consume 300 g of mashed potatoes.
  Arms: Canola oil only / 10 min preload (All 24 participants)

SUMMARY:
The objective of this study is to investigate the importance of leavy vegetable preloading on the postprandial glycaemic and insulinemic response in human subjects when consumed a specific amount of digestible carbohydrate from Russet Burbank potatoes source.

DETAILED DESCRIPTION:
The proposed research is part of strategies to manipulate postprandial glycemia and generate weight-control-related benefits, such as promoting satiation. Literature has shown pre-loading caloric nutrients can change postprandial glycemia, but the mechanism is unclear. The investigators hypothesize that a small number of nutrients released in the small intestine can initiate physiological changes and develop feedback control to delay gastric emptying, leading to the delay in digestion of glycemic carbohydrates and the consequent moderate glycemic responses. The investigators propose to use potatoes as the testing glycemic carbohydrates, and the pre-load foods are green vegetables. The investigators will be testing the optimal preload time to achieve the highest control of glycemic response as well as the strongest effect in satiety induction. In addition, green vegetables will be consumed with or without a preload fat enhancer (canola oil) to investigate the mechanism behind significant preload compositions. Healthy adults will be instructed to eat the leafy vegetables first (with or without canola oil), followed by the potato foods (i.e., mashed potatoes). The measurement is the gastric emptying time, blood sugar concentration, insulin, and an appetite-related gut hormone GLP-1. In order to monitor gastric emptying using a non-invasive approach, a popular breath test used in children and a hydrogen breath test will be used to present the change of gastric emptying and the level of gut fermentation.

Results will demonstrate the mechanism of the impact of pre-loading nutrients on the digestion of glycemic carbohydrates. The goal is to eliminate the negative influence of glycemic carbohydrate consumption. Instead, to generate health benefits from dietary carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (18.5 kg/m2 to 24.9 kg/m2), weight >/= 45 kg
* Normal blood pressure </=120/80 mmH
* Fasting blood glucose of <5.6 mmol/l
* Able to provide written informed consent before participating in the study.
* Able to communicate adequately to comply with the requirements of the entire study, i.e., able to eat test meal and provide breath samples.

Exclusion Criteria:

* Smokers.
* Individuals with any metabolic diseases (such as diabetes, hypertension etc).
* Individuals with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency).
* Individuals with medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics).
* Individuals who take any prescribed medication or dietary supplements which may interfere with the study measurements.
* Individuals who have any major organ dysfunction (eg. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug.
* Individuals with history of malabsorption due to mucosal disease, pancreatic disease, or other causes.
* Individuals with history of gastrointestinal disease or surgery (excludes appendectomy, hernia repair and anorectal disorders).
* Individuals who are allergic/intolerant to any of the test foods to be administered, or any of the following common food and ingredients: eggs, fish, milk, peanuts, tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, sulphites etc.
* People who intentionally restrict food intake.
* People who consume excessive 13C rich products such as corn, sugar beet and pineapple.
* Individuals who partake in sports at the competitive and/or endurance levels
* Individuals who have any known chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV).
* Individuals who is a study team member or an immediate family of any study team member.
* Individuals who consume Excessive alcohol: consuming >/= 6 alcoholic drinks per week.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood glucose | up to 3 hour (180 minutes) after test meal consumption
  Blood samples are taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 minutes. Glucose levels are tested in the serum using cobas c311 analyzer.
Postprandial blood Insulin | up to 3 hour (180 minutes) after test meal consumption
  Blood samples are taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 minutes. Insulin levels are tested in the serum using cobas e411 Immunoanalyzer.
Postprandial Glucagon Like Peptide -1 Total (GLP-1) | up to 3 hour (180 minutes) after test meal consumption
  Blood samples are taken at baseline, 15, 30, 45, 60, 90, 120, 150 and 180 minutes. GLP-1 levels are tested in the plasma using GLP-1 Total ELISA kit (EZGLP1T-36K)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lin, PhD, Principal Investigator — Senior Principal Scientist I at Singapore Institute of Food and Biotechnology Innovation
Locations (1):
- Clinical Nutrition Research Centre (CNRC), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
According to the approved IRB# 2021-095, all IPD are owned by Singapore Institute of Food and Biotechnology Innovation (SIFBI)